CLINICAL TRIAL: NCT03735160
Title: Monitoring the Pressure Over Nasotracheal Intubation and Related Nasal Alar Injury
Brief Title: Pressure Over Nasotracheal Intubation Related Nasal Alar Injury
Status: Withdrawn | Type: Observational
Why Stopped: Technical problem
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chien-Chung,Huang, Principal Investigator,Attending physician of anesthesiology, Mackay Memorial Hospital
Other Study IDs: 18MMHIS084e
Record Dates: First submitted 2018-11-06; First posted 2018-11-08 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Intubation Complication; Pressure Injury
Keywords: Nasotracheal intubation; nasal alar injury
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nasal intubation with pressure sensor: anesthetized patient with nasotracheal intubation
  Interventions: Device: pressure sensor

INTERVENTIONS:
Device: pressure sensor — Pressure sensor at the angle of intratracheal tube and nasal alar

SUMMARY:
Nasotracheal intubation can cause injury and hemorrhage of nasal mucosa and nasal alar. The investigators measure the actual pressure at the angle between nasotracheal tube and nasal alar, analyze the relationship of clinical signs and symptoms to build up optimal clinical routines.

DETAILED DESCRIPTION:
While assisting ventilation during general anesthesia or other reasons, patients are often intubated with endotracheal tube to secure airway. Endotracheal tube can be placed trans-orally or trans-nasally according to surgical conditions, anatomical considerations and nursing needs. Except inadequate cuff pressure related complication, nasotracheal intubation can cause dysfunction of nasal mucosal cilia, injury and hemorrhage of nasal mucosa, turbinate avulsion, obstruction of nasal airway, sinusitis and compression and injury of nasal alar, resulting in local erythema, ischemia, pressure sore, necrosis, tissue damage and may affect appearance.

Previous studies focus on the process of nasal tracheal intubation, aim to reduce mucosal injury and hemorrhage via specific intubation tool, special endotracheal tube design, lubricant and so on. However, evidences in preventing nasal alar injury are limited, in which injuries are mostly prevented by self-made special endotracheal tube and artificial leather. In general, the etiology of tissue damage is compression pressure exceeding local capillary perfusion pressure, resulting in reduced perfusion, ischemia and necrosis. Clinically, health providers prevent the injury by standardized endotracheal tube fixation and/or artificial leather at sites with potential compression. But the extend of the effect of endotracheal tube to trachea mucosa varies, range of pressure affecting capillary perfusion pressure are not yet defined, and no routine monitoring for dermis compression. Thus, endotracheal tube related skin damage is an important clinical issue without best standard operating procedure.

In this study, the investigators will place a pressure sensor at the angle of nasotracheal tube, measure the actual pressure, define the sites of compression and its pressure, analyze the relationship of clinical signs and symptoms, pressure, and duration of nasotracheal intubation, and build up optimal clinical routines.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Physical classification I & II
* patients undergo general anesthesia and receive intratracheal intubation through nose
* elective surgery

Exclusion Criteria:

* with known nasal injury
* already intubation before induction
* surgery on the nose
* emergent operation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergo general anesthesia and receive intratracheal intubation through nose
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
appearance of nose | from induction to one day after surgery
  intact or redness ; if redness then, go through NPUAP classification
VAS | from induction to one day after surgery
  Patient's VISUAL ANALOG SCALE (VAS) for pain of the nose after surgery: no pain (0 - 4 mm), mild pain (5- 44mm), moderate pain (45-74 mm), and severe pain (75-100 mm)
pressure between nose and intratracheal tube | during intubation
  pressure between nose and intratracheal tube detected by pressure sensors
NPUAP classification | from induction to one day after surgery
  The National Pressure Ulcer Advisory Panel stage

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Chung Huang, MD, Study Director — Mackay Memorial Hospital
Locations (1):
- MacKay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Seegobin RD, van Hasselt GL. Endotracheal cuff pressure and tracheal mucosal blood flow: endoscopic study of effects of four large volume cuffs. Br Med J (Clin Res Ed). 1984 Mar 31;288(6422):965-8. doi: 10.1136/bmj.288.6422.965. PMID 6423162
- [Result] Schneider J, Mulale U, Yamout S, Pollard S, Silver P. Impact of monitoring endotracheal tube cuff leak pressure on postextubation stridor in children. J Crit Care. 2016 Dec;36:173-177. doi: 10.1016/j.jcrc.2016.06.033. Epub 2016 Jul 9. PMID 27546768
- [Result] Al-Metwalli RR, Sadek S. Safety and reliability of the sealing cuff pressure of the Microcuff pediatric tracheal tube for prevention of post-extubation morbidity in children: A comparative study. Saudi J Anaesth. 2014 Oct;8(4):484-8. doi: 10.4103/1658-354X.140856. PMID 25422605
- [Result] Bolzan DW, Gomes WJ, Peixoto TC, Faresin SM, Carvalho AC, De Paola AA, Guizilini S. Clinical use of the volume-time curve for endotracheal tube cuff management. Respir Care. 2014 Nov;59(11):1628-35. doi: 10.4187/respcare.02683. Epub 2014 Jun 10. PMID 24917452
- [Result] Bernhard WN, Cottrell JE, Sivakumaran C, Patel K, Yost L, Turndorf H. Adjustment of intracuff pressure to prevent aspiration. Anesthesiology. 1979 Apr;50(4):363-6. doi: 10.1097/00000542-197904000-00018. No abstract available. PMID 434545
- [Result] Elwany S, Mekhamer A. Effect of nasotracheal intubation on nasal mucociliary clearance. Br J Anaesth. 1987 Jun;59(6):755-9. doi: 10.1093/bja/59.6.755. PMID 3606919
- [Result] Neves-Pinto RM, Carvalho A, Araujo E, Alberto C, Basilio-De-Oliveira, De Carvalho GA. Nasal septum giant pyogenic granuloma after a long lasting nasal intubation: case report. Rhinology. 2005 Mar;43(1):66-9. PMID 15844505
- [Result] Holzapfel L. Nasal vs oral intubation. Minerva Anestesiol. 2003 May;69(5):348-52. PMID 12768165
- [Result] Kuo MJ, Reid AP, Smith JE. Unilateral nasal obstruction: an unusual presentation of a complication of nasotracheal intubation. J Laryngol Otol. 1994 Nov;108(11):991-2. doi: 10.1017/s0022215100128701. PMID 7829957
- [Result] Yeom JH, Oh MK, Shin WJ, Ahn DW, Jeon WJ, Cho SY. Randomized comparison of the effectiveness of nasal intubation using a GlideScope video laryngoscope with Magill forceps versus vascular forceps in patients with a normal airway. Can J Anaesth. 2017 Dec;64(12):1176-1181. doi: 10.1007/s12630-017-0971-4. Epub 2017 Sep 26. PMID 28952139
- [Result] Sanuki T, Hirokane M, Matsuda Y, Sugioka S, Kotani J. The Parker Flex-Tip tube for nasotracheal intubation: the influence on nasal mucosal trauma. Anaesthesia. 2010 Jan;65(1):8-11. doi: 10.1111/j.1365-2044.2009.06123.x. Epub 2009 Oct 22. PMID 19849677
- [Result] Song J. A comparison of the effects of epinephrine and xylometazoline in decreasing nasal bleeding during nasotracheal intubation. J Dent Anesth Pain Med. 2017 Dec;17(4):281-287. doi: 10.17245/jdapm.2017.17.4.281. Epub 2017 Dec 28. PMID 29349350
- [Result] Cherng CH, Chen YW. Using a modified nasotracheal tube to prevent nasal ala pressure sore during prolonged nasotracheal intubation. J Anesth. 2010 Dec;24(6):959-61. doi: 10.1007/s00540-010-1009-z. Epub 2010 Sep 1. PMID 20809246
- [Result] Huang TT, Tseng CE, Lee TM, Yeh JY, Lai YY. Preventing pressure sores of the nasal ala after nasotracheal tube intubation: from animal model to clinical application. J Oral Maxillofac Surg. 2009 Mar;67(3):543-51. doi: 10.1016/j.joms.2008.06.100. PMID 19231778
- [Result] Meier R, Sporn P. [Decubitus ulcer prevention in the nasal ala using Silastic foam in nasotracheal intubated patients]. Anaesthesist. 1986 Jan;35(1):49-50. German. PMID 3963354